CLINICAL TRIAL: NCT03906786
Title: Motivational Interviewing and Self-care in Type 1 Diabetes: Randomized Controlled Clinical Trial.
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Hospital Universitario Insular Gran Canaria (Other)
Collaborators: Menarini Group (Industry)
Responsible Party: Principal Investigator, Rosa María Sánchez Hernández, Clinical Doctor, Hospital Universitario Insular Gran Canaria
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: CEIm-CHUIMI-2017/974
Record Dates: First submitted 2019-03-25; First posted 2019-04-08 (Actual); Last update posted 2019-04-08 (Actual); Status verified 2019-04

CONDITIONS: Type1diabetes
Keywords: self-care; motivational interviewing; doctor-pacient relationship
MeSH Terms: interventions — Motivational Interviewing

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- motivacional interviewing group (Experimental)
  Interventions: Behavioral: motivational interviewing
- control group (No Intervention)

INTERVENTIONS:
Behavioral: motivational interviewing — The intervention will consist of 4 structured medical consultations in the form of a motivational interviewing compared to usual care, covering a 12-month intervention period. In both groups, the frequency of visits (c / 3 months) and the variables collected will be the same.
  Arms: motivacional interviewing group

SUMMARY:
Type 1 diabetes requires a high level of involvement of patients to obtain good control by following complex therapeutic recommendations. Motivational Interviewing has proven to be effective in changing behaviors in sedentary people, with addictions and with obesity.

Our objective is to evaluate the impact of an intervention with Motivational Interviewing in patients with type 1 diabetes, through a randomized controlled clinical trial. At least sixty patients with type 1 diabetes will be included with HbA1c> 8% that will be randomized with a ratio of 1: 1. In the intervention group, Motivational Interviewing will be applied in the routine clinical appointments with the Endocrinologist, while the control group will receive the same visits but in a traditional way.

The primary result will be self-care behaviors according to a validated questionnaire. Secondary outcomes include: HbA1c, number of hypoglycemia, motivation with self-care, self-efficacy, quality of life, compliance with patients' own objectives, lipid profile, weight and blood pressure.

The professionals will be trained in Motivational Interviewing with the objective of favoring the adherence to self-care, the motivation of the patient and improving doctor-patient relationship. They will also be evaluated through a specific questionnaire.

ELIGIBILITY:
Inclusion Criteria:

* Patients with DM1 seen in outpatient clinics of Endocrinology and Nutrition with at least one year of evolution, HbA1c> 8% and / or severe hypoglycemia in the previous 6 months

Exclusion Criteria:

* Gestion underway or scheduled for the next 9 months. Any circumstance that, in the opinion of the investigators, could interfere with the follow-up of the patient.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 60 (Estimated)
Dates: Start 2019-03-07 (Actual); Primary Completion 2020-09-30 (Estimated); Study Completion 2020-09-30 (Estimated)

PRIMARY OUTCOMES:
Adherence to self-care behaviors. The Diabetes Self-Care Inventory-Revised | 12 months
  The validated Spanish version of The Diabetes Self-Care Inventory-Revised version (SCI-R) (18) was used. This inventory consists of 15 items that refer to self-care behaviors in the treatment of diabetes, which are scored on a Likert scale ranging from (1 = "never" to 5 = "always"). The scores are converted with a formula and the responses range from 0-100; higher scores indicate higher levels of self-care

CONTACTS AND LOCATIONS:
Overall Officials: Ana M Wägner, Principal Investigator — Hospital Universitario Insular de Gran Canaria
Locations (1):
- Complejo Hospitalario Universitario Materno-infantil de Las Palmas, Las Palmas de Gran Canaria, Las Palmas, Spain

IPD SHARING:
Plan to Share IPD: Yes
Anonimized results will be available upon request
Supporting Information: Study Protocol, SAP
Time Frame: Protocol and statistical plan: as son as posible Access to results. Upon publication
Access Criteria: Study protocol and statistical analysis plan will be published (draft in progress) Individual data/results (anonimized) will be available upon request

REFERENCES:
- [Derived] Alvarado-Martel D, Boronat M, Alberiche-Ruano MDP, Algara-Gonzalez MA, Ramallo-Farina Y, Wagner AM. Motivational Interviewing and Self-Care in Type 1 Diabetes: A Randomized Controlled Clinical Trial Study Protocol. Front Endocrinol (Lausanne). 2020 Dec 10;11:574312. doi: 10.3389/fendo.2020.574312. eCollection 2020. PMID 33362714